CLINICAL TRIAL: NCT02110329
Title: Simultaneous Detection of Somatic Quantitative Molecular Alterations Using the Qantitative Multiplex Pcr of Short Fluorescent Fragments Method (QMPSF) in Stage II-III Colon Cancer: a Prospective Study
Brief Title: Simultaneaous Detection of Quantitative Somatic Alterations Using the Qantitative Multiplex Pcr of Short Fluorescent Fragments Method (QMPSF) in Stage II-III Colon Cancer: a Prospective Study
Acronym: Code Barre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2007/040/HP
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer; Stage II and III
Keywords: colorectal cancer; stage II and III; somatic quantitative molecular alterations; Qantitative Multiplex Pcr of Short fluorescent Fragments method (QMPSF)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- stage II-III colon cancer treated with surgery (No Intervention): stage II-III colon cancer treated with surgery
  Interventions: Genetic: evaluation of the recurrence rate according to molecular analysis

INTERVENTIONS:
Genetic: evaluation of the recurrence rate according to molecular analysis

SUMMARY:
Lymph node involvement remains the main criteria for postoperative chemotherapy in patients with colon cancer (CC) without distant metastasis. To date, the prognostic value of the somatic quantitative molecular alterations such as loss or gain of genomic region is not established in CC.

AIMS & METHODS: Using the one-step screening method based on the Quantitative Multiplex PCR of Short fluorescent Fragments (QMPSF), we aimed to assess the prognostic role of the simultaneous detection of main quantitative somatic alterations in stage II-III CC.

Patients and Methods. We enrolled and collected all baseline characteristics of patients operated for a stage II-III CC with storage frozen tissues. The QMPSF was based on a simultaneous amplification of 9 selected target genomic sequences from literature: DCC (18q21); EGFR (7p12); P53 (17p13.1); BLK (8p23-p22); c-myc (8q24.12); APC (5q22.2); ERBB2 (17q12); STK6 (20q13.31); NR21 (14p11.1) and two control: DCOHM (5q31.1); HMBS (11q23.3). Comparison of each amplicon electropherograms obtained from tumour vs normal peritumoral tissue allowed us to identified gain or loss genomic region. The primary end-point was the local and/or distant recurrence and relation between clinical and single or combined molecular alterations and recurrence were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* localized colon cancer
* proven adenocarcinoma
* surgery R0
* no metastatic disease
* stage II or III
* WHO performance status 0, 1 or 2
* availaible frozen tissue
* written consent
* no major co-morbidities

Exclusion Criteria:

* metastatic disease
* hereditary colorectal cancer
* rectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Recurence rate according to molecular results | 36 months
  Using the one-step screening method based on the Quantitative Multiplex PCR of Short fluorescent Fragments (QMPSF), we aimed to assess the prognostic role of the simultaneous detection of main quantitative somatic alterations in stage II-III CC.

SECONDARY OUTCOMES:
Survival rate according to molecular results | 60 months
  Using the one-step screening method based on the Quantitative Multiplex PCR of Short fluorescent Fragments (QMPSF), we aimed to assess the prognostic role of the simultaneous detection of main quantitative somatic alterations in stage II-III CC.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Dijon, Dijon
  - Chu Lille, Lille
  - Chu Hopitaux de Rouen, Rouen